CLINICAL TRIAL: NCT01301014
Title: Reliability and Diagnostic Accuracy of an Alternate Lachman's Test Performed in a Prone Position
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ed Mulligan, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: ProneLachman1
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2011-02

CONDITIONS: Anterior Cruciate Ligament Stability
Keywords: accuracy, anterior cruciate ligament, diagnostic value, examination, knee, Lachman test, sensitivity, specificity
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is investigating the reliability and diagnostic accuracy of a Lachman's test conducted in a prone position to detect the presence of a torn anterior cruciate ligament.

ELIGIBILITY:
Inclusion Criteria:

* current knee pain complaint in subjects between 15 and 60 years old

Exclusion Criteria:

* the inability to assume the prone testing position
* evidence of a fracture by application of the Ottawa Fracture rule
* previous knee joint arthroplasty
* suspicion of posterior cruciate involvement
* knee surgery in the previous six months
* presence of serious underlying non-mechanical pathology
* systemic illness

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 31 men and 21 women ranging in age from 16-57 years old with complaint of knee pain
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Mulligan EP, Harwell JL, Robertson WJ. Reliability and diagnostic accuracy of the Lachman test performed in a prone position. J Orthop Sports Phys Ther. 2011 Oct;41(10):749-57. doi: 10.2519/jospt.2011.3761. Epub 2011 Sep 4. PMID 21891874